CLINICAL TRIAL: NCT03481114
Title: Patient-Reported Outcomes Following Chemoradiotherapy for Locally Advanced Non-small Cell Lung Cancer: A Randomized Trial Comparing Two Radiotherapy Schedules
Brief Title: Patient-Reported Outcomes Following Chemoradiotherapy for Locally Advanced Non-small Cell Lung Cancer
Acronym: REPAINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8065
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: radiation therapy; chemotherapy; PET Imaging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard chemoradiotherapy (Active Comparator): Patients receiving standard radiotherapy will receive a total dose of 60 Gy in 30 fractions over 6 weeks, delivered to all involved lesions (tumors and lymph nodes).
  Interventions: Combination Product: Standard chemoradiotherapy
- PET-based, dose-painted, accelerated chemoradiotherapy, (Experimental): For patients receiving PET-based, dose-painted, accelerated chemoradiotherapy, lesions with MTV exceeding 20 cc will be treated with 55 Gy in 20 fractions over 4 weeks, while lesions with MTV below 20 cc will receive 44 Gy in 20 fractions over the same 4 weeks.
  Interventions: Combination Product: PET-based, dose-painted, accelerated chemoradiotherapy

INTERVENTIONS:
Combination Product: PET-based, dose-painted, accelerated chemoradiotherapy — Patients in this arm will receive a more personalized and shorter radiation therapy treatment course utilizing PET imaging.
  Arms: PET-based, dose-painted, accelerated chemoradiotherapy,
Combination Product: Standard chemoradiotherapy — Patients in this arm will receive a standard radiotherapy course.
  Arms: Standard chemoradiotherapy

SUMMARY:
The primary objective of this study is to evaluate patient-reported outcomes during and after concurrent chemoradiotherapy for locally-advanced non-small cell lung cancer. Patients will be randomized to a standard 6-week radiotherapy course or a 4-week radiotherapy course using dose-painting based on pre-treatment PET findings.

DETAILED DESCRIPTION:
This study is open for patients with non-small cell lung cancer. This study offers such patients the chance for a shorter and more personalized treatment course utilizing PET imaging.

Patients will be stratified based on performance status and tumor size and randomized to one of two treatment plans:

1. PET-based, dose-painted, accelerated chemoradiotherapy over 4 weeks (20 radiotherapy fractions)
2. Standard chemoradiotherapy over 6 weeks (30 radiotherapy fractions)

All patients will receive standard weekly doses of chemotherapy (carboplatin and paclitaxel) during radiotherapy. This may be followed by adjuvant systemic therapy, at the discretion of the treating physicians.

All patients will undergo standard evaluations prior to enrollment, during treatment, and after treatment. Additionally, patient-reported outcomes will be assessed periodically using a PRO-CTCAE tool.

ELIGIBILITY:
Inclusion Criteria:

Pathologically proven (either histologic or cytologic) diagnosis of NSCLC with any of the following stages (according to the AJCC Staging Manual, 7th edition,

Appendix):

* Stage IIIA or IIIB
* Stage II NSCLC with contraindication to curative surgical resection
* Stage IV disease with solitary brain metastasis that has been treated radically (eg: with surgical resection and/or stereotactic radiosurgery) and thoracic disease that would be classified as stage II-III

Appropriate diagnostic/staging workup, including:

* Complete history and physical examination
* PET/CT within 42 days prior to study entry demonstrating hypermetabolic pulmonary lesion(s) and/or thoracic lymph node(s). If PET/CT was obtained more than 42 days prior to study entry and is not repeated, chest CT within 28 days prior to study entry demonstrating stable disease is required.
* MRI of the brain or head CT with contrast within 42 days prior to study entry
* No prior chemotherapy or thoracic radiotherapy for lung cancer
* ECOG Performance Status 0-2
* Age > 18
* Able to read and write in one of the following languages, in which the PROCTCAE tool is available: English, Danish, German, Italian, Japanese, Korean, Spanish
* Laboratory studies obtained within 28 days prior to study entry demonstrating adequate bone marrow and end organ function
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of study therapy, agree to utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study therapy is completed,and be advised of the importance of avoiding pregnancy during trial participation and the potential risks of an unintentional pregnancy.

All patients must sign study specific informed consent prior to study entry.

Exclusion Criteria:

* Pleural or pericardial effusion (A patient with pleural effusion may be enrolled the effusion is sampled by thoracentesis and cytology is negative or the effusion is seen on axial imaging but not on chest x-ray and deemed too small to tap under CT or ultrasound guidance.)
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
* Women who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study therapy
* have a positive pregnancy test at baseline
* are pregnant or breastfeeding
* Poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) despite attempts to improve glucose control by fasting duration and adjustment of medications. Patients with diabetes will preferably be scheduled for PET/CT imaging in the morning, and instructions for fasting and use of medications will be provided in consultation with the patients' primary physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
PRO-CTCAE adverse events with score ≥ 3, observed 6 weeks after initiation of chemoradiotherapy | 6 Weeks after initiation of Chemoradiation

SECONDARY OUTCOMES:
Locoregional progression-free survival | Weeks 19, 32 and 45 on study
  Lack of local disease progression based on repeat imaging
Progression-free survival | Weeks 19, 32 and 45 on study
  Lack of any disease progression based on repeat imaging
Overall survival | From treatment start through 5 years post treatment
  Follow ups will be maintained with study patients to determine survival status
Grade 3-5 adverse events, scored using CTCAE v. 4 | From treatment start through study week 45
  Evaluation of any side effects or toxicities using a standard grading system
PRO-CTCAE adverse events with score ≥ 3 at any time | From treatment start through study week 45
  Evaluation of severe, patient reported side effects or toxicities
PRO-CTCAE adverse events with any score | From treatment start through study week 45
  Evaluation of any patient reported side effects or toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No